CLINICAL TRIAL: NCT06254417
Title: Study of Diaphragmatic Ultrasound as a Predictor of Mechanical Ventilation in Patients With Respiratory Diseases on Admission to Intensive Care Unit
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, RAMY AHMED, Assistant Professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: master ICU
Record Dates: First submitted 2024-01-28; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Respiratory Disease
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NON VENTILATED GROUP (Active Comparator)
  Interventions: Procedure: Diaphragmatic ultrasound
- VENTILATED GROUP (Active Comparator)
  Interventions: Procedure: Diaphragmatic ultrasound

INTERVENTIONS:
Procedure: Diaphragmatic ultrasound — Diaphragmatic ultrasound will be performed to all patients with respiratory disease to evaluate diaphragmatic thickening and estimate thickening fraction and to evaluate diaphragmatic excursion. Measurements will be obtained at bedside with a portable ultrasound machine equipped with a linear probe (Logic P6 Pro, GE Healthcare). Diaphragmatic thickness measures will be performed on right Intercostal approach through the zone of apposition. Diaphragmatic excursion will be performed using curved-array probe (Logic P6 Pro, GE Healthcare) is positioned below right costal arch at the mid-clavicular line. The ultrasound study will be done and /or supervised by ultrasound expert

SUMMARY:
Ultrasonography has been used to explore diaphragmatic contractile activity by measuring thickening fraction .When thickening fraction was < 20% during tidal breathing, it is commonly associated with respiratory failure.

Diaphragmatic ultrasound had been used before as a tool to predict weaning from mechanical ventilation.

In this study diaphragmatic ultrasound will be done upon admission to predict of mechanical ventilation in patients with respiratory diseases.

DETAILED DESCRIPTION:
All Patients will be subjected to the following Detailed history taking from patient or relatives including the cause of respiratory diseases.

Complete physical examination: general and local examination will be carried out for all patients.

All cases undergo standard monitoring including invasive and non-invasive blood pressure monitoring, SpO2 and ECG.

Full laboratory investigations: At the beginning of the study (Arterial blood gases, CBC, Coagulation Profile, Kidney function tests, Liver function tests, Cardiac enzymes).

All patients will be treated according to the international guidelines according to their medical status . As well as Hemodynamic support will be provided by fluids resuscitation and/or catecholamine infusion if necessary, to keep mean arterial pressure >70 mmHg.

Respiratory support will consist of oxygen administration or mechanical ventilation if necessary, to maintain SPO2 > 90% and PH > 7.25.

Diaphragmatic ultrasound will be performed to all patients with respiratory disease to evaluate diaphragmatic thickening and estimate thickening fraction and to evaluate diaphragmatic excursion. Measurements will be obtained at bedside with a portable ultrasound machine equipped with a linear probe (Logic P6 Pro, GE Healthcare). Diaphragmatic thickness measures will be performed on right Intercostal approach through the zone of apposition. Diaphragmatic excursion will be performed using curved-array probe (Logic P6 Pro, GE Healthcare) is positioned below right costal arch at the mid-clavicular line. The ultrasound study will be done and /or supervised by ultrasound expert.

The decision of using mechanical ventilation will not depend on the diaphragmatic ultrasound results.

Primary outcome: estimation of diaphragmatic thickening fraction which will predict mechanical ventilation.

Secondary outcome: estimation of diaphragmatic excursion which will predict mechanical ventilation.

Non invasive ventilation (NIV) will be delivered through a full-face mask connected to a high-performance ventilator. In non-invasive pressure support mode. PEEP and delivered FIO2 will be set to achieve oxygen saturation target of 88-92%. Pressure support level will be adjusted to obtain a target volume of 6-8 mL/kg, a frequency < 30 breaths/min, and air leak < 15%. Cycling will be set at 40% of peak flow. If non-invasive ventilation failed or patient deteriorated invasive ventilation will be required.

Indication of non invasive ventilation:

* Moderate to sever dyspnea increased over usual , respiratory rate more than24 cycle/ min, accessory muscle use and paradoxical breathing.
* Pao2 more than 55 mmHg.
* PH between 7.25 and 7.35.
* Pao2 /Fio2 less than 200.
* Hypoxia So2 less than 88% on O2

Indication of invasive ventilation:

* any contraindication of non invasive ventilation.
* Failure of non invasive ventilation after (1:2) hours.
* Hemodynamic instability. (Decrease base line values >20% on admission)

ELIGIBILITY:
Inclusion Criteria:

* Dyspnea: respiratory rate > 22 breaths per min.
* Hypoxia: as SO2 < 92% on room air.
* Hypercapnia: as PaCO2 > 45mmHg.

Exclusion Criteria:

* Age <18 year.
* Cardiogenic pulmonary edema.
* History of interstitial lung disease (fibrosis).
* Neuromuscular disease.
* Significant chest wall deformities.
* Previous diagnosis of diaphragmatic palsy.
* Recent thoracotomy or sternotomy (within the previous year).
* Severe hemodynamic instability or shock.
* Pregnancy.
* Diagnosis of pneumothorax or pneumo mediastinum.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
estimation of diaphragmatic thickening fraction | immediately after intensive care admission

SECONDARY OUTCOMES:
estimation of diaphragmatic excursion | immediately after intensive care admission
  measurement of the movement of the diaphragm during breathing by ultrasonography(normally about 3-5 centimeter)